CLINICAL TRIAL: NCT05579730
Title: Evaluation of Combination Drug Product Brimonidine Tartrate 0.025%/Ketotifen Fumarate 0.035% Ophthalmic Solution Compared to Its Components and Vehicle for the Treatment of Allergic Conjunctivitis in the Conjunctival Allergen Challenge Model
Brief Title: Evaluation of Brimonidine Tartrate/Ketotifen Fumarate Combination for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 909
Record Dates: First submitted 2022-10-06; First posted 2022-10-14 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Combination (Experimental): Brimonidine tartrate 0.025%/ketotifen fumarate 0.035% combination ophthalmic solution
  Interventions: Drug: Brimonidine tartrate 0.025%/ketotifen fumarate 0.035%
- Ketotifen fumarate (Active Comparator): ketotifen fumarate 0.035% ophthalmic solution
  Interventions: Drug: Ketotifen Fumarate 0.035%
- Brimonidine tartrate (Active Comparator): brimonidine tartrate 0.025% ophthalmic solution
  Interventions: Drug: Brimonidine Tartrate 0.025%
- Vehicle (Placebo Comparator): vehicle ophthalmic solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Brimonidine tartrate 0.025%/ketotifen fumarate 0.035% — combination ophthalmic solution
  Arms: Combination
Drug: Brimonidine Tartrate 0.025% — ophthalmic Solution
  Arms: Brimonidine tartrate
Drug: Ketotifen Fumarate 0.035% — ophthalmic Solution
  Arms: Ketotifen fumarate
Drug: Vehicle — ophthalmic Solution
  Arms: Vehicle

SUMMARY:
To evaluate the efficacy of Combo (Drug Product Brimonidine Tartrate 0.025%/Ketotifen Fumarate 0.035% Ophthalmic Solution) compared to its individual components and vehicle in a population of subjects with allergic conjunctivitis:

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  1. be at least 10 years of age of either sex and any race;
  2. provide written informed consent and sign a HIPAA form. Subjects who are under the age of 18 will need to sign an assent form as well as having a parent or legal guardian sign an informed consent;
  3. be willing and able to follow all instructions and attend all study visits;
  4. (If female and of childbearing potential) agree to have urine pregnancy testing performed at visits 2, 4a (must be negative) and at exit visit (Visit 5); must not be lactating; and must agree to use at least 1 medically acceptable form of birth control throughout the study duration, for at least 14 days prior to the first dose of investigational drug (Visit 4a) and for 1 month after the last dose of investigational drug (Visit 5). Acceptable forms of birth control are true abstinence (when this is in line with the preferred and usual lifestyle of the subject), spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of male partner at least 3 months prior to the first dose of investigational drug (Visit 4a). Note: Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
  5. (If male and with female partner of childbearing potential) must use at least 1 medically acceptable form of birth control. throughout the study duration, for at least 14 days prior to the first dose of investigational drug (Visit 4a) and for 1 month after the last dose of the study drug (Visit 5) Note: Acceptable forms of birth control are true abstinence (when this is in line with the preferred and usual lifestyle of the subject) or vasectomy at least 3 months prior to the first dose of investigational drug (Visit 4a). Without a vasectomy, must use condoms with spermicidal foam/gel/film/cream/suppository.
  6. have a history of ocular allergies and a positive skin test reaction to a seasonal (grass, ragweed, tree pollen) or perennial (cat dander, dog dander, dust mites, cockroach) allergen as confirmed by an allergic skin test conducted at Visit 1 or within the past 24 months;
  7. have a calculated best-corrected visual acuity of 0.7 LogMar or better in each eye as measured using an ETDRS chart at Visit 2;
  8. have a positive bilateral CAC reaction (defined as having scores of ≥ 2 for ocular itching and ≥ 2 for conjunctival redness) within 10 minutes of instillation of the last titration of allergen at Visit 2;
  9. have a positive bilateral CAC reaction (defined as having scores of ≥ 2 for ocular itching and ≥ 2 for conjunctival redness) in at least 2 out of 3 timepoints at following the challenge at Visit 3;
  10. be able and willing to discontinue wearing contact lenses for at least 72 hours prior to Visit 2 and during the study trial period.

Exclusion Criteria:

* Subjects may not:

  1. have known contraindications or sensitivities to the use of any of the investigational product(s) or their components;
  2. have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters (including but not limited to narrow angle glaucoma, clinically significant blepharitis, follicular conjunctivitis, iritis, pterygium, or a diagnosis of dry eye);
  3. have had ocular surgical intervention within 3 months prior to enrollment (Visit 4a) and/or a history of refractive surgery within 6 months prior to enrollment (Visit 4a);
  4. have a known history of retinal detachment, diabetic retinopathy, or progressive retinal disease;
  5. have the presence of an active ocular infection (bacterial, viral or fungal), positive history of an ocular herpetic infection, or preauricular lymphadenopathy at any visit;
  6. manifest signs or symptoms of clinically active allergic conjunctivitis in either eye at the start of Visits 2, 3, or 4a (defined as a score of >0 for itching and/or >1 for conjunctival redness);
  7. use any of the following disallowed medications during the period indicated prior to Visit 2 and agree not to use disallowed medications throughout the study:

  7 Days
  * systemic or ocular H1 antihistamines, H1 antihistamine/mast-cell stabilizer drug combinations, H1 antihistamine-vasoconstrictor drug combinations,
  * decongestants,
  * immunotherapeutic agents,
  * monoamine oxidase inhibitors,
  * artificial tears,
  * eye whiteners (eg, vasoconstrictors),
  * lid scrubs,
  * mast cell stabilizers,
  * prostaglandins or prostaglandin derivatives,
  * ocular, topical, or systemic nonsteroidal anti-inflammatory drugs (NSAIDs);

    *Baby aspirin (81 mg) is allowed as long as a stable dose has been maintained for at least 30 days prior to Visit 1 and will continue to be maintained for the duration of the study.

    14 Days
  * inhaled, ocular, topical, or systemic corticosteroids or mast cellstabilizers;

    45 Days
  * depo-corticosteroids

    2 Months
  * immunosuppressive or cancer chemotherapeutic agents

Note: Currently marketed over-the counter anti-allergy eyedrops (i.e., antihistamine/vasoconstrictor combination products like Visine-A®or Naphcon-A®) may be administered to subjects at the end of each visit, after all evaluations are completed;

8. have any significant illness (for example, any autoimmune disease requiring therapy, or severe cardiovascular disease [including arrhythmias]) the Investigator feels could be expected to interfere with the subject's safety or study parameters and/or put the subject at any unnecessary risk (includes but is not limited to poorly controlled hypertension or poorly controlled diabetes, a history of status asthmaticus, organ transplants, a known history of persistent moderate or severe asthma, or a known history of moderate to severe allergic asthmatic reactions to any of the study allergens);

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - 103, Phoenix, Arizona
  - 101, Andover, Massachusetts
  - 102, Memphis, Tennessee
  - 114, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination: Brimonidine tartrate 0.025% / ketotifen fumarate 0.035% combination ophthalmic solution administered bilaterally.
- Ketotifen Fumarate: Ketotifen fumarate ophthalmic solution 0.035% administered bilaterally
- Brimonidine Tartrate: Brimonidine tartrate ophthalmic solution 0.025% administered bilaterally
- Vehicle: Vehicle ophthalmic solution administered bilaterally
Period: Overall Study
Arm/Group | Combination | Ketotifen Fumarate | Brimonidine Tartrate | Vehicle
Started | 47 | 48 | 47 | 46
Completed | 45 | 45 | 47 | 44
Not Completed | 2 | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Combination: Brimonidine tartrate 0.025% / ketotifen fumarate 0.035% ophthalmic solution administered bilaterally
- Total: Total of all reporting groups
Arm/Group | Combination | Ketotifen Fumarate | Brimonidine Tartrate | Vehicle | Total
Number analyzed (Participants) | 47 | 48 | 47 | 46 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (16.90) | 49.3 (14.19) | 45.9 (17.74) | 49.9 (12.18) | 48.1 (15.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 32 | 26 | 122
  Male | 13 | 18 | 15 | 20 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 6 | 2 | 18
  Not Hispanic or Latino | 42 | 43 | 41 | 44 | 170
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching
Description: Ocular itching score (measured on a 0-4 unit scale, allowing half-unit increments; average score of the subject's two eyes) assessed by the subjects at 3 (±1), 5 (±1), and 7 (±1) minutes post-CAC.
Time Frame: Assessed at Visit 4b on day 1 (duration of action CAC at 8 hours post-instillation of study medication) and Visit 5 on day 15 (onset of action CAC at 15 minutes post-instillation of study medication).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Combination | Ketotifen Fumarate | Brimonidine Tartrate | Vehicle
Number analyzed (Participants) | 47 | 48 | 47 | 46
score on a scale
  Visit 4b, 3 min Post-CAC | 1.176 (0.1464) | 1.708 (0.1487) | 2.426 (0.1330) | 2.362 (0.1512)
  Visit 4b, 5 min Post-CAC | 1.287 (0.1507) | 1.688 (0.1519) | 2.638 (0.1155) | 2.712 (0.1427)
  Visit 4b, 7 min Post-CAC | 1.181 (0.1462) | 1.656 (0.1532) | 2.644 (0.1249) | 2.755 (0.1390)
  Visit 5, 3 min Post-CAC | 0.495 (0.0918) | 0.594 (0.1296) | 1.915 (0.1307) | 2.070 (0.1319)
  Visit 5, 5 min Post-CAC | 0.601 (0.0930) | 0.791 (0.1350) | 1.973 (0.1255) | 2.345 (0.1378)
  Visit 5, 7 min Post-CAC | 0.618 (0.1083) | 0.972 (0.1548) | 1.920 (0.1394) | 2.358 (0.1221)

2. Primary Outcome: Conjunctival Redness
Description: Conjunctival redness score (measured on a 0-4unit scale, allowing half-unit increments; average score of the subject's two eyes) assessed by investigator at 7 (±1), 15 (±1), and 20 (±1) minutes post-CAC.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Combination | Ketotifen Fumarate | Brimonidine Tartrate | Vehicle
Number analyzed (Participants) | 47 | 48 | 47 | 46
score on a scale
  Visit 4b, 7 min Post-CAC | 1.372 (0.1088) | 1.844 (0.0895) | 1.883 (0.1083) | 2.155 (0.0850)
  Visit 4b, 15 min Post-CAC | 1.617 (0.1204) | 2.130 (0.0939) | 2.069 (0.1189) | 2.321 (0.0934)
  Visit 4b, 20 min Post-CAC | 1.649 (0.1165) | 2.146 (0.0953) | 1.984 (0.1296) | 2.315 (0.0961)
  Visit 5, 7 min Post-CAC | 0.591 (0.0846) | 1.393 (0.0944) | 1.005 (0.1300) | 2.052 (0.1143)
  Visit 5, 15 min Post-CAC | 0.765 (0.1043) | 1.662 (0.1036) | 1.069 (0.1338) | 2.268 (0.1111)
  Visit 5, 20 min Post-CAC | 0.735 (0.1012) | 1.727 (0.1088) | 1.021 (0.1343) | 2.238 (0.1182)

ADVERSE EVENTS:
Time Frame: Assessed through the study, approximately 10 weeks
Arm/Group | Combination | Ketotifen Fumarate | Brimonidine Tartrate | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48 | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48 | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 3/47 | 6/48 | 6/47 | 4/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination (N=47) | Ketotifen Fumarate (N=48) | Brimonidine Tartrate (N=47) | Vehicle (N=46)
Visual Acuity reduced (Eye disorders) | 1 | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Instillation site foreign body sensation (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT05579730/Prot_002.pdf
  • Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT05579730/SAP_003.pdf